CLINICAL TRIAL: NCT04835220
Title: Trial of Oral Lenalidomide Stewardship Program for Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: W.G. Bill Hefner Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Goodman, Principal Investigator, W.G. Bill Hefner Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-42
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Medication Compliance
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Telehealth intervention group and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Electronic pill bottle cap (MEMs bottle cap) with no Telehealth calls
- Telehealth intervention group (Other): Electronic pill bottle cap (MEMs bottle cap) with regular telehealth visits to the veterans at the VAMCs on the stewardship program. These visits will involve contacting the veterans by telephone, administering a questionnaire to review their medication-taking behavior for oral chemotherapy, and potentially contacting the treating oncologist in the event that the veterans are at risk of non-adherence (based on their responses).
  Interventions: Other: Telehealth Calls

INTERVENTIONS:
Other: Telehealth Calls — The telehealth nurse will record data in a case report form within the VA REDCap electronic data capture system that is stored within the VA firewall.
  Arms: Telehealth intervention group

SUMMARY:
To address the challenge of oral chemotherapy stewardship in the Veteran population, this study outlines the implementation and evaluation of a pilot program for the delivery and management of lenalidomide to increase the adherence rates. Our goal is to utilize a team-based multi-disciplinary approach using existing technological resources such as the tele-oncology program at the Salisbury VA and other VA medical centers to provide cancer care that is safe, effective, compassionate, and cost-effective. Subject will be prescribed a Lenalidomide based therapy per standard of care. Eligibility is based only on a prescription for Lenalidomide and is independent of any other concurrent treatments for myeloma. The objectives are as followed: 1. To describe the demographics and baseline clinical characteristics of veterans with newly diagnosed multiple myeloma treated with oral lenalidomide. 2. To evaluate the impact of the stewardship program (intervention) on the adherence to oral lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with myeloma or Initiating lenalidomide maintenance therapy after transplant or transplant ineligible patients that are started on lenalidomide until progression or intolerance.
* Myeloma diagnosis (International Classification of Diseases, Tenth Revision, Clinical Modification [ICD-10-CM] codes:vC90.00 or associated diagnosis )
* Prescription for lenalidomide
* Planned or Currently treated with lenalidomide as part of a treatment regimen for newly diagnosed myeloma
* Renal function assessed by calculated creatinine clearance as follows (see Appendix: Cockcroft-Gault estimation of CrCl):

Subjects must have calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula. (See Appendix C). Dosing for patients with creatinine clearance between 30ml/min-60ml/min will be based on lenalidomide package insert.

* Total bilirubin 1.5 x ULN
* AST (SGOT) and ALT (SGPT) 3 x ULN.
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Able to take prophylactic anticoagulation such as aspirin, warfarin, low molecular weight heparin or direct oral anticoagulant.
* Personal Computer with internet Capability.

Exclusion Criteria:

* < 18 years of age as of the index date
* Newly diagnosed with myeloma and not started on lenalidomide
* Known hypersensitivity to thalidomide or lenalidomide (if applicable).
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Females who are pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2024-03-26 (Estimated); Study Completion 2024-03-26 (Estimated)

PRIMARY OUTCOMES:
Adherence of medication compliance | 12 Months
  To evaluate the impact of the stewardship program (intervention) on the adherence to oral lenalidomide. Adherence of veterans to their prescribed lenalidomide treatment will be measured based on MEMs bottle cap data. A descriptive analysis using data from the MGL Scale (asked during the telehealth call) will be conducted to describe adherence in the stewardship assistance program cohort. Of note, patients in the intervention arm who stop attending telehealth calls prior to the completion of the patient stewardship program will still be considered as part of the intervention arm (i.e., an "intent-to-treat analysis"). However, data on the participation in the patient stewardship program (e.g., number of telehealth visits attended), will be collected and may be used in sensitivity analyses if appropriate.

SECONDARY OUTCOMES:
Clinical Characteristics | 12 months
  Describe the demographics and baseline clinical characteristics of veterans with newly diagnosed multiple myeloma treated with oral lenalidomide.

CONTACTS AND LOCATIONS:
Locations (1):
- W.G. Bill Hefner VAMC, Salisbury, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No